CLINICAL TRIAL: NCT04931108
Title: The Effect of Nitrendipine/Atenolol Combination on Blood Pressure Variability of Patients With Grade 1 Hypertension Compared With Nitrendipine or Atenolol Monotherapy.
Brief Title: The Effect of Nitrendipine/Atenolol Combination on Blood Pressure Variability.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NAC-BPV
Record Dates: First submitted 2021-05-27; First posted 2021-06-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
Keywords: blood pressure variability; nitrendipine; atenolol
MeSH Terms: conditions — Hypertension | interventions — Nitrendipine; Atenolol

STUDY DESIGN:
Intervention Model Description: Half of patients will take nitrendipine/atenolol (5/10mg) once daily for 6 weeks first, and then evenly turn into nitrendipine (10mg) or atenolol (25mg) once daily for 6 weeks. Another half of patients will evenly take nitrendipine (10mg) or atenolol (25mg) first, and turn into nitrendipine/atenolol (5/10mg) next.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): One pill of nitrendipine/atenolol combination (5/10mg) once daily for 6 weeks first, and followed by monotherapy for another 6 weeks, when patients will evenly assigned to one pill of nitrendipine (10mg) or one pill of atenolol (25mg) once daily.
  Interventions: Drug: Nitrendipine/Atenolol; Drug: Nitrendipine; Drug: Atenolol
- Sequence 2 (Experimental): Monotherapy for 6 weeks first, when patients will evenly assigned to one pill of nitrendipine (10mg) or one pill of atenolol (25mg) once daily, followed by one pill of nitrendipine/atenolol combination (5/10mg) once daily for another 6 weeks.
  Interventions: Drug: Nitrendipine/Atenolol; Drug: Nitrendipine; Drug: Atenolol

INTERVENTIONS:
Drug: Nitrendipine/Atenolol — Nitrendipine/Atenolol 5mg/10mg single-pill combination, oral tablet, one pill daily.
  Other Names: Nitrendipine and Atenolol Tablets
Drug: Nitrendipine — Nitrendipine 5mg, oral tablet, one pill daily.
  Other Names: Nitrendipine Tablets
Drug: Atenolol — Atenolol 25mg, oral tablet, one pill daily.
  Other Names: Atenolol Tablets

SUMMARY:
1. Study name: The Effect of Nitrendipine/Atenolol Combination on Blood Pressure Variability.
2. Medicine: Nitrendipine/Atenolol; Nitrendipine; Atenolol.
3. Rationale: Blood pressure variability correlates with cardiovascular events and target-organ damage in hypertensive patients. Nitrendipine/Atenolol has obvious advantages in reducing blood pressure variability in hypertensive rats, but the effect of this combination on hypertensive patients is still unknown.
4. Objective: To evaluate the effect of nitrendipine/atenolol on blood pressure variability of patients with Grade 1 hypertension compared with nitrendipine or atenolol monotherapy.
5. Study design: This study is a cross-over, randomized, controlled clinical trial with two equally sized treatment groups: Nitrendipine/Atenolol (5mg/10mg); Nitrendipine (10mg) or atenolol (25mg).
6. Study population: Men and Women aged 30-65 years (n=32) meeting the inclusion/exclusion criteria.
7. Randomization and cross-over design: Eligible patients will be randomly divided into two groups. Half of patients will take nitrendipine/atenolol (5/10mg) once daily for 6 weeks first, and then evenly turn into nitrendipine (10mg) or atenolol (25mg) once daily for 6 weeks. Another half of patients will evenly take nitrendipine (10mg) or atenolol (25mg) first, and turn into nitrendipine/atenolol (5/10mg) next.
8. Follow up: 14 weeks.
9. Sample size: a total of 32 patients should be enrolled.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in April 2021, recruitment will start. Patients enrollment and follow-up will be performed between June 2021 to June 2022.

DETAILED DESCRIPTION:
1. Study name: The effect of Nitrendipine/Atenolol combination on blood pressure variability of patients with Grade 1 hypertension compared with nitrendipine or atenolol monotherapy.
2. Medicine: Nitrendipine/Atenolol (5/10mg tablet); Nitrendipine (10mg tablet); Atenolol (25mg tablet)
3. Rationale: Blood pressure variability correlates with cardiovascular events and target-organ damage in hypertensive patients. Nitrendipine/Atenolol has obvious advantages in reducing blood pressure variability in hypertensive rats, but the effect of this combination on hypertensive patients is still unknown.
4. Objective: To evaluate the effect of nitrendipine/atenolol on blood pressure variability of patients with Grade 1 hypertension compared with nitrendipine or atenolol monotherapy.
5. Study design: This study is a cross-over, randomized, controlled clinical trial with two equally sized treatment groups: Nitrendipine/Atenolol (5mg/10mg); Nitrendipine (10mg) or atenolol (25mg).
6. Study population: Eligible patients (n=32) should be men or women aged 30-65 years. Untreated patients diagnosed as essential hypertension, whose daytime systolic blood pressure ≥ 135mmHg and/or daytime diastolic blood pressure ≥ 85mmHg, and standard deviation (SD)≥13mmHg will be recruited.
7. Randomization and cross-over design: Eligible patients will be randomly divided into two groups. Half of patients will take nitrendipine/atenolol (5/10mg) once daily for 6 weeks first, and then evenly turn into nitrendipine (10mg) or atenolol (25mg) once daily for 6 weeks. Another half of patients will evenly take nitrendipine (10mg) or atenolol (25mg) first, and turn into nitrendipine/atenolol (5/10mg) next.
8. Follow up: 14 weeks. 1 week for screening period, 6 weeks for the first period of treatment, 1 week for wash-out period, and 6 weeks for the second period of treatment.
9. Sample size: a total of 32 patients should be enrolled.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in April 2021, recruitment will start. Patients enrollment and follow-up will be performed between June 2021 to June 2022.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women.
* Aged 30-65 years.
* Ambulatory systolic blood pressure ≥ 135 mmHg and/or diastolic blood pressure ≥ 85 mmHg.
* Ambulatory daytime systolic blood pressure standard deviation (SD)≥13mmHg.
* Never took antihypertensive drugs.
* Signed the written consent.

Exclusion Criteria:

* Under antihypertensive treatments.
* Clinic systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg.
* Contraindications to the treatment of drugs, including hypersensitivity reaction, bradycardia, asthma, etc.
* Any cardiovascular disease except hypertension.
* Suspected or confirmed secondary hypertension.
* Poor compliance.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Ambulatory systolic blood pressure variability 1 | The first 6 weeks of treatment.
  Including the average real variability (ARV), the coefficient of variation (CV),and the standard deviation (SD).
Ambulatory systolic blood pressure variability 2 | The second 6 weeks of cross-over treatment.
  Including the average real variability (ARV), the coefficient of variation (CV),and the standard deviation (SD).

SECONDARY OUTCOMES:
Ambulatory diastolic blood pressure variability 1 | The first 6 weeks of treatment.
  Including the average real variability (ARV), the coefficient of variation (CV),and the standard deviation (SD).
Ambulatory diastolic blood pressure variability 2 | The second 6 weeks of cross-over treatment.
  Including the average real variability (ARV), the coefficient of variation (CV),and the standard deviation (SD).
Ambulatory blood pressure 1 | The first 6 weeks of treatment.
  Including ambulatory blood pressure over 24 hours, daytime and nighttime.
Ambulatory blood pressure 2 | The second 6 weeks of cross-over treatment.
  Including ambulatory blood pressure over 24 hours, daytime and nighttime.

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xia JH, Cheng YB, Xu TY, Guo QH, Chan CM, Hu LX, Li Y, Wang JG. Effect of a calcium-channel blocker and beta-blocker combination on reading-to-reading blood pressure variability: a randomized crossover trial. Blood Press Monit. 2025 Apr 1;30(2):73-81. doi: 10.1097/MBP.0000000000000736. Epub 2024 Nov 26. PMID 39831760